CLINICAL TRIAL: NCT04735484
Title: Measuring Dynamic Spinal Balance With Wearable Activity Trackers. A Case Control Study.
Brief Title: Spinal Balance With Wearables - Case-control
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University College, London (Other)
Collaborators: Royal National Orthopaedic Hospital NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: EDGE132844
Record Dates: First submitted 2021-01-28; First posted 2021-02-03 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-01

CONDITIONS: Adolescent Idiopathic Scoliosis
MeSH Terms: interventions — Gait Analysis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (2):
- Case: Participants will attend one data collection appointment wearing form-fitting sports clothing and trainers. Participants will wear infrared markers and wearable devices whilst walking over level ground and on a treadmill. Data will be collected using a motion capture system and the wearable devices themselves. Data collection will take approximately 90 minutes
  Interventions: Device: Gait analysis
- Control: Participants will attend one data collection appointment wearing form-fitting sports clothing and trainers. Participants will wear infrared markers and wearable devices whilst walking over level ground and on a treadmill. Data will be collected using a motion capture system and the wearable devices themselves. Data collection will take approximately 90 minutes
  Interventions: Device: Gait analysis

INTERVENTIONS:
Device: Gait analysis — Collecting movement data whilst participants walk

SUMMARY:
Observational case-control study to see if the Margin of Stability and Dynamic Postural Stability (measured using a motion capture gait laboratory and wearable device, respectively) are different in children with Adolescent Idiopathic Scoliosis and matched controls. Participants will walk across level ground and on a treadmill once for data collection and no follow-up is required.

DETAILED DESCRIPTION:
The goal of this observational case-control study is to validate the Margin of Stability (MoS) and Dynamic Postural Stability (DPS) measures using a motion capture gait laboratory and wearable device in patients with Adolescent Idiopathic Scoliosis (AIS).

These measures will provide a consultant with objective data about a patient's movement and balance that the consultant and other healthcare professionals can use to infer about their spinal deformity progression or improvement. This research is an early step for working towards providing a distance medicine, non-invasive outcome measure that can be used alongside or in the absence of current clinical measures and radiography. Use of this data could reduce the frequency with which radiographs are required and so reduce the impact of radiation exposure. This wearable device could complement and improve upon existing outcome measures in the treatment of spinal deformity, reduce the need for radiographs and ameliorate the need for distance patient monitoring methods. A motion capture gait laboratory will be used as the gold-standard comparison.

A pilot study has been carried out on healthy participants with a simulated spinal deformity in a kinematic gait laboratory and using the wearable device, which showed altered balance in the simulated scoliosis group compared to controls.

The aim of this project is to:

1. To see if there's a difference in MoS and DPS between children with AIS and controls,
2. To see if a difference can be detected using motion capture gait analysis and a wearable device,
3. To see how similar results from the wearable device are to the motion capture gait laboratory,
4. To test the ability of the wearable device to measure a scalable difference between radiographic curve magnitude in patients with AIS.

Participants will attend one data collection appointment where they will walk across level ground and on a treadmill. No follow-up is required.

ELIGIBILITY:
Case Inclusion Criteria:

* Diagnosed with Adolescent Idiopathic Scoliosis
* Single, right-sided thoracic, left-sided thoraco-lumbar or left-sided lumbar curve
* <= 1cm leg length discrepancy
* Diagnostic radiographs of curvature within 3 months
* Ability to walk without assistance
* Willing and able to comply with clinical study visit requirements

Control Inclusion Criteria:

* Ability to walk without assistance
* Willing and able to comply with clinical study visit requirements

Case & Control Exclusion Criteria:

* Previous spinal surgery or joint replacement
* Syndromic, neuromuscular or pathologic condition
* Neurological, vestibular, somatosensory or orthopaedic comorbidities
* Pregnancy
* Poor understanding of written and/or spoken English

Ages: 10 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patient records will be accessed by a member of the clinical care team with legitimate access to patient records and who is independent to the research team to identify eligible patients as 'Case' participants. These patients and their parents will be approached with a letter asking them to contact the researcher if they are interested in participating. Additionally, recruitment posters will be displayed in the RNOH outpatient and RNOH orthotics departments.
  For 'Control' participants, with permission from the participating schools and colleges, a letter will be sent to parents of children aged 10-18 at local schools and colleges requesting they volunteer for this study.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2021-05 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Margin of stability | Data collection appointment 1 - approx. 90 minutes

SECONDARY OUTCOMES:
Dynamic Postural Stability | Data collection appointment 1 - approx. 90 minutes
Correlation between Margin of Stability and radiographic Cobb angle | Data collection appointment 1 - approx. 90 minutes
Correlation between Dynamic Postural Stability and radiographic Cobb angle | Data collection appointment 1 - approx. 90 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Rui Loureiro, Principal Investigator — University College, London

IPD SHARING:
Plan to Share IPD: Undecided